CLINICAL TRIAL: NCT03003962
Title: A Phase III Randomized, Open-Label, Multi-Center Study of Durvalumab (MEDI4736) Versus Standard of Care (SoC) Platinum-Based Chemotherapy as First Line Treatment in Patients With PD-L1-High Expression Advanced Non Small-Cell Lung Cancer
Brief Title: Study of Durvalumab Alone or Chemotherapy for Patients With Advanced Non Small-Cell Lung Cancer (PEARL)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419AC00002; 2018-001375-21 (EudraCT Number)
Record Dates: First submitted 2016-12-15; First posted 2016-12-28 (Estimated); Results first posted 2023-12-26 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Carcinoma NSCLC
Keywords: NSCLC; PD-L1; Durvalumab (MEDI4736); OS
MeSH Terms: interventions — durvalumab; CP protocol; Gemcitabine; Cisplatin; Carboplatin; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: Durvalumab (Experimental): Anti-PD-L1 monoclonal Antibody monotherapy
  Interventions: Drug: Durvalumab (MEDI4736)
- Arm 2: Standard of Care (Active Comparator): Standard of Care Platinum-Based chemotherapy
  Interventions: Drug: Paclitaxel + carboplatin; Drug: Gemcitabine + cisplatin; Drug: Gemcitabine + carboplatin; Drug: Pemetrexed + cisplatin; Drug: Pemetrexed + carboplatin

INTERVENTIONS:
Drug: Durvalumab (MEDI4736) — Anti-PD-L1 monoclonal Antibody monotherapy
  Arms: Arm 1: Durvalumab
Drug: Paclitaxel + carboplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Arm 2: Standard of Care
Drug: Gemcitabine + cisplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Arm 2: Standard of Care
Drug: Gemcitabine + carboplatin — Chemotherapy Agents
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Arm 2: Standard of Care
Drug: Pemetrexed + cisplatin — Chemotherapy Agent
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Arm 2: Standard of Care
Drug: Pemetrexed + carboplatin — Chemotherapy Agent
  Other Names: Platinum based Standard of Care Chemotherapy
  Arms: Arm 2: Standard of Care

SUMMARY:
This is a randomized, open-label, multi-center Phase III study to determine the efficacy and safety of durvalumab versus platinum-based SoC chemotherapy in the first-line treatment of advanced NSCLC in patients who are epidermal growth factor receptor (EGFR) and anaplastic lymphoma kinase (ALK) wild-type and with PD-L1 high expression (PEARL)

DETAILED DESCRIPTION:
Patients with stage IV NSCLC will be randomized in a 1:1 ratio to 2 treatment arms (durvalumab or SOC therapy). The dual primary objectives of this study are to assess the efficacy of durvalumab versus SoC in terms of OS (Overall Survival) in all randomized patients and in patients who are at low risk of EM (early mortality)

ELIGIBILITY:
Inclusion Criteria

* Aged at least 18 years
* Documented evidence of Stage IV NSCLC
* No sensitizing EGFR mutation and ALK rearrangement
* PD-L1 high expression
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion Criteria:

* Prior chemotherapy or any other systemic therapy for advanced NSCLC
* Prior exposure to immune-mediated therapy, including, but not limited to, other anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4), anti-programmed cell death1 (PD-1), anti-programmed cell death ligand 1 (PD-L1), or anti PD-L2 antibodies, excluding therapeutic anticancer vaccines
* Brain metastases or spinal cord compression unless the patient is stable and off steroids for at least 14 days prior to start of study treatment
* Mixed small-cell lung cancer and NSCLC histology, sarcomatoid variant
* Active or prior documented autoimmune or inflammatory disorders (e.g., colitis or Crohn's disease]

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2022-10-27 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Locations (69):
- Research Site, Anaheim, California, United States
- Australia (4):
  - Research Site, Box Hill
  - Research Site, Gosford
  - Research Site, Kogarah
  - Research Site, St Leonards
- China (24):
  - Research Site, Beijing
  - Research Site, Bengbu
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Jinan
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shijiazhuang
  - Research Site, Ürümqi
  - Research Site, Wanzhou
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
  - Research Site, Zhuhai
- Hungary (6):
  - Research Site, Budapest
  - Research Site, Deszk
  - Research Site, Farkasgyepü
  - Research Site, Gyöngyös - Mátraháza
  - Research Site, Székesfehérvár
  - Research Site, Törökbálint
- Research Site, Almelo, Netherlands
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Grudziądz
  - Research Site, Koszalin
  - Research Site, Lublin
  - Research Site, Mrozy
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (7):
  - Research Site, Arkhangelsk
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Omsk
  - Research Site, Rostov-on-Don
  - Research Site, Saint Petersburg
  - Research Site, Volgograd
- South Korea (7):
  - Research Site, Changwon-si
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Incheon
  - Research Site, Jinju
  - Research Site, Seoul
  - Research Site, Suwon
- Taiwan (2):
  - Research Site, Taichung
  - Research Site, Taipei
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Muang
  - Research Site, Songkhla
- Turkey (Türkiye) (4):
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Malatya
  - Research Site, Pamukkale
- Vietnam (3):
  - Research Site, Can Tho
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419AC00002&attachmentIdentifier=78e650f3-53a9-42f0-8ee7-98654cae7412&fileName=d419ac00002_CSR_Synopsis.pdf&versionIdentifier=
- See also: CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419AC00002&attachmentIdentifier=e22a0ee4-f267-4a3e-8427-8d623ae5b200&fileName=D419AC00002_Protocol.pdf&versionIdentifier=
- See also: SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D419AC00002&attachmentIdentifier=32bffb61-41f6-4de8-9d93-66b17672af32&fileName=d419ac00002_SAP.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase III, open-label, multi-center study was conducted in participants with programmed cell death ligand 1 (PD-L1)- tumor cell (TC) >= 25% advanced non small-cell lung cancer (NSCLC) at 85 centers in 10 countries (China, Russia, Hungary, Poland, South Korea, Vietnam, Turkey, Australia, Taiwan, and Thailand). First participant was enrolled on 02 January 2017 and last participant was enrolled on 25 January 2019.
Pre-assignment Details: Overall 3075 participants were screened at 98 centers in 12 countries. A total of 669 participants were randomized in a 1:1 ratio. Of those, 549 participants fulfilled the criteria for PD-L1 TC >= 25% low risk of early mortality (LREM).
Groups:
- Durvalumab: Participants received durvalumab 20 milligram (mg)/kilogram (kg) via intravenous (IV) infusion every 4 weeks (Q4W) until documented disease progression (PD) or unacceptable toxicity or until specific treatment discontinuation criteria were met.
- Platinum-based SoC: Participants received 1 of the following IV infusion treatment combination platinum-based standard of care (SoC) as per Investigator's choice on Day 1 of each 21-day cycle for 4 to 6 cycles or until documented PD or until specific treatment discontinuation criteria were met.
  1. Paclitaxel 175 mg/ square meter (m^2) and carboplatin area under the plasma concentration curve (AUC) 5 or 6 via IV infusions.
  2. Gemcitabine 1000 or 1250 mg/m^2 and cisplatin 75 or 80 mg/m^2 (for squamous participants).
  3. Gemcitabine 1000 or 1250 mg/m^2 and carboplatin AUC 5 or 6 via infusions (for squamous participants).
  4. Pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 (for non-squamous participants; pemetrexed maintenance dose was permitted).
  5. Pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6 via IV infusions (for non-squamous participants; pemetrexed maintenance dose was permitted).
Period: Overall Study
Arm/Group | Durvalumab | Platinum-based SoC
Started (Randomized) | 335 | 334
PD L1 TC ≥ 25% LREM Analysis Set | 278 | 271
PD L1 TC ≥ 50% Analysis Set | 247 | 246
PD L1 TC ≥ 50% LREM Analysis Set | 207 | 199
Completed | 1 | 0
Not Completed | 334 | 334
Not completed — Withdrawal by Subject | 5 | 17
Not completed — Death | 274 | 277
Not completed — Participants ongoing at DCO | 55 | 40

BASELINE CHARACTERISTICS:
Population: The Full analysis set (FAS) included all randomized participants.
Groups:
- Durvalumab: Participants received durvalumab 20 mg/kg via IV infusion Q4W until documented PD or unacceptable toxicity or until specific treatment discontinuation criteria were met.
- Platinum-based SoC: Participants received 1 of the following IV infusion treatment combination platinum-based SoC as per Investigator's choice on Day 1 of each 21-day cycle for 4 to 6 cycles or until documented PD or until specific treatment discontinuation criteria were met.
  1. Paclitaxel 175 mg/m^2 and carboplatin AUC 5 or 6 via IV infusions.
  2. Gemcitabine 1000 or 1250 mg/m^2 and cisplatin 75 or 80 mg/m^2 (for squamous participants).
  3. Gemcitabine 1000 or 1250 mg/m^2 and carboplatin AUC 5 or 6 via infusions (for squamous participants).
  4. Pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 (for non-squamous participants; pemetrexed maintenance dose was permitted).
  5. Pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6 via IV infusions (for non-squamous participants; pemetrexed maintenance dose was permitted).
- Total: Total of all reporting groups
Arm/Group | Durvalumab | Platinum-based SoC | Total
Number analyzed (Participants) | 335 | 334 | 669
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.7 (9.73) | 61.9 (8.71) | 61.3 (9.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 65 | 132
  Male | 268 | 269 | 537
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 73 | 61 | 134
  Asian | 262 | 273 | 535
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 6 | 8
  Not Hispanic or Latino | 333 | 328 | 661

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of randomization until death due to any cause (date of death or censoring-date of randomization + 1). Any participant not known to have died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive.
Time Frame: From date of randomization until death due to any cause. Assessed up to a maximum of approximately 69 months [data cut-off (DCO) 27 October 2022]
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 335 | 334
months | 14.6 [12.2 to 16.9] | 12.8 [10.1 to 14.7]
Statistical Analysis 1: Comparison: Durvalumab vs Platinum-based SoC; Test type: Other — The analysis was performed using the stratified log-rank test, adjusting for PD-L1 expression (TC 25% to 49% versus >= 50%) and histology and smoking status (squamous vs. non-squamous + never smoker vs. non-squamous + former/current smoker) and using the rank tests of association approach; p = 0.037, Stratified Log-rank test; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.706 to 0.989] — The HR and confidence interval (CI) were calculated using a stratified Cox proportional hazards model

2. Primary Outcome: OS in Participants With LREM
Description: as for outcome 1
Time Frame: From date of randomization until death due to any cause. Assessed up to a maximum of approximately 69 months (DCO 27 October 2022)
Population: The PD-L1 TC >= 25% LREM analysis set included participants identified by a prognostic model developed by AstraZeneca as having LREM.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 278 | 271
months | 14.6 [12.6 to 17.2] | 15.0 [13.1 to 16.8]
Statistical Analysis 1: Comparison: Durvalumab vs Platinum-based SoC; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.628, Stratified log-rank test; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.793 to 1.151] — The HR and CI were calculated using a stratified Cox proportional hazards model

3. Secondary Outcome: OS in PD-L1 TC >= 50% Analysis Set
Description: as for outcome 1
Time Frame: as for outcome 2
Population: The PD-L1 TC >= 50% analysis set included the subset of participants in the FAS whose PD-L1 expression status was PD-L1 TC >= 50% as defined by the VENTANA PD-L1 (SP263) assay.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 247 | 246
months | 14.6 [12.0 to 17.7] | 11.8 [9.8 to 14.7]

4. Secondary Outcome: OS in PD-L1 TC >= 50% LREM Analysis Set
Description: OS is defined as the time from the date of randomization until death due to ay cause (date of death or censoring-date of randomization + 1). Any participant not known to have died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive.
Time Frame: as for outcome 2
Population: The PD-L1 TC >= 50% LREM analysis set included participants with PD-L1 TC >= 50% and identified by a prognostic model developed by AstraZeneca as having LREM.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Platinum-based SoC: Participants received 1 of the following IV infusion treatment combination platinum-based SoC as per Investigator's choice on Day 1 of each 21-day cycle for 4 to 6 cycles or until documented PD or until specific treatment discontinuation criteria were met.
  1. Paclitaxel 175 mg/m^2 and carboplatin AUC 5 o 6 via IV infusions.
  2. Gemcitabine 1000 or 1250 mg/m^2 and cisplatin 75 or 80 mg/m^2 (for squamous participants).
  3. Gemcitabine 1000 or 1250 mg/m^2 and carboplatin AUC 5 or 6 via infusions (for squamous participants).
  4. Pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 (for non-squamous participants; pemetrexed maintenance dose was permitted).
  5. Pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6 via IV infusions (for non-squamous participants; pemetrexed maintenance dose was permitted).
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 207 | 199
months | 14.9 [12.6 to 19.0] | 14.9 [11.8 to 17.7]

5. Secondary Outcome: Progression Free Survival (PFS) Based on Investigator Assessment According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: The PFS (per RECIST 1.1) was defined as the time from the date of randomization until the date of objective disease progression or death regardless of whether the participants withdrew from randomized therapy or received another anticancer therapy prior to progression (i.e., date of PFS event or censoring - date of randomization +1). Progression of disease per RECIST 1.1, when either 1 of the criteria met: Target lesion (TL): at least a 20% increase in the sum of diameters of TLs, for reference the smallest sum on study. In addition, the sum must also demonstrate an absolute increase of at least 5 millimeters (mm). Non-target lesion (NTL): Unequivocal progression of existing NTLs. It may be due to an important progression in 1 lesion only or in several lesions. In all cases the progression must be clinically significant for the physician to consider changing (or stopping) therapy. New lesions: the presence of 1 or more new lesions was assessed as progression.
Time Frame: Tumor assessments (per RECIST 1.1) every 6 weeks for the first 48 weeks relative to the date of randomization and then every 8 weeks thereafter until confirmed objective disease progression (up to a maximum of approximately 69 months DCO 27 October 2022)
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 335 | 334
months | 5.4 [4.2 to 5.7] | 4.8 [4.3 to 5.6]

6. Secondary Outcome: PFS Based on Investigator Assessment According to RECIST 1.1 in LREM Analysis Set
Description: The PFS (per RECIST 1.1 using Investigator assessments) was defined as the time from the date of randomization until the date of objective disease progression or death regardless of whether the participants withdrew from randomized therapy or received another anticancer therapy prior to progression (i.e., date of PFS event or censoring - date of randomization +1).
Time Frame: Tumor assessments (per RECIST 1.1) every 6 weeks for the first 48 weeks relative to the date of randomization and then every 8 weeks thereafter until confirmed objective disease progression (up to a maximum of approximately 69 months)
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 278 | 271
months | 5.5 [4.4 to 6.4] | 5.6 [4.8 to 5.9]

7. Secondary Outcome: PFS Based on Investigator Assessment According to RECIST 1.1 in PD-L1 TC >= 50% Analysis Set
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 247 | 246
months | 5.6 [4.7 to 6.5] | 4.5 [4.2 to 5.6]

8. Secondary Outcome: PFS Based on Investigator Assessment According to RECIST 1.1 in PD-L1 TC >= 50% LREM Analysis Set
Description: as for outcome 6
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 207 | 199
months | 5.7 [5.3 to 7.0] | 5.5 [4.2 to 5.7]

9. Secondary Outcome: Objective Response Rate (ORR) as Per RECIST 1.1 Using Investigator Assessment
Description: ORR (per RECIST 1.1 using Investigator assessments) was defined as the percentage of participants with an unconfirmed response of complete response (CR) or partial response (PR). CR was defined as disappearance of all target lesions (TLs). Any pathological lymph nodes selected as TLs had a reduction in short axis to < 10 millimeter (mm). PR was defined as at least a 30% decrease in the sum of diameters of TLs, with reference the baseline sum of diameters if criteria for PD are not met.
Time Frame: as for outcome 6
Population: The FAS included all randomized participants who had PD-L1 expression TC >= 25% with the VENTANA PD-L1 (SP263) assay.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 335 | 334
percentage of participants | 37.6 [0.324 to 0.430] | 37.4 [0.322 to 0.429]

10. Secondary Outcome: ORR as Per RECIST 1.1 Using Investigator Assessment in PD-L1 TC >= 25% LREM Analysis Set
Description: ORR (per RECIST 1.1 using Investigator assessments)was defined as the percentage of participants with an unconfirmed response of CR or PR. CR was defined as disappearance of all TLs. Any pathological lymph nodes selected as TLs had a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of TLs, with reference the baseline sum of diameters if criteria for PD are not met.
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 278 | 271
percentage of participants | 38.5 [0.327 to 0.445] | 40.2 [0.343 to 0.463]

11. Secondary Outcome: ORR as Per RECIST 1.1 Using Investigator Assessment in PD-L1 TC >= 50% Analysis Set
Description: ORR (per RECIST 1.1 using Investigator assessments) was defined as the percentage of participants with an unconfirmed response of CR or PR. CR was defined as disappearance of all TLs. Any pathological lymph nodes selected as TLs had a reduction in short axis to < 10 mm. PR was defined as at least a 30% decrease in the sum of diameters of TLs, with reference the baseline sum of diameters if criteria for PD are not met.
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 247 | 246
percentage of participants | 42.1 [0.359 to 0.485] | 40.7 [0.345 to 0.471]

12. Secondary Outcome: ORR as Per RECIST 1.1 Using Investigator Assessment in PD-L1 TC >= 50% LREM Analysis Set
Description: as for outcome 11
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 207 | 199
percentage of participants | 44.0 [0.371 to 0.510] | 43.7 [0.367 to 0.509]

13. Secondary Outcome: Duration of Response (DoR) as Per RECIST 1.1 Using Investigator Assessment
Description: DoR (per RECIST 1.1 using Investigator assessments) was defined as the time from the date of first documented response until the first date of documented progression or death in the absence of disease progression (i.e. date of PFS event or censoring - date of first response + 1). DoR was calculated using the Kaplan-Meier technique.
Time Frame: as for outcome 6
Population: The FAS included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 126 | 125
months | 11.9 [9.7 to 18.7] | 4.2 [3.3 to 4.6]

14. Secondary Outcome: DoR as Per RECIST 1.1 Using Investigator Assessment in PD-L1 TC >=25% LREM Analysis Set
Description: as for outcome 13
Time Frame: as for outcome 6
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 107 | 109
months | 11.6 [8.2 to 15.7] | 4.2 [4.0 to 5.4]

15. Secondary Outcome: DoR as Per RECIST 1.1 Using Investigator Assessment in PD-L1 TC >=50% Analysis Set
Description: as for outcome 13
Time Frame: as for outcome 6
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 104 | 100
months | 12.2 [8.3 to 21.2] | 4.2 [3.0 to 4.6]

16. Secondary Outcome: DoR as Per RECIST 1.1 Using Investigator Assessment in PD-L1 TC >=50% LREM Analysis Set
Description: as for outcome 13
Time Frame: as for outcome 6
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 91 | 87
months | 12.2 [8.2 to 19.7] | 4.2 [3.9 to 5.4]

17. Secondary Outcome: Alive and Progression-Free at 12 Months (APF12)
Description: The APF12 was defined as the Kaplan-Meier estimate of percentage of participants alive and progression free at 12 months based on PFS (per RECIST 1.1 as assessed using Investigator assessments) analysis.
Time Frame: From date of randomization until 12 months
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 335 | 334
percentage of participants | 25.5 [20.8 to 30.4] | 13.3 [9.6 to 17.5]

18. Secondary Outcome: APF12 in PD-L1 TC >= 25% LREM Analysis Set
Description: as for outcome 17
Time Frame: From date of randomization until 12 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 278 | 271
percentage of participants | 24.1 [19.1 to 29.5] | 16.4 [11.9 to 21.5]

19. Secondary Outcome: APF12 in PD-L1 TC >= 50% Analysis Set
Description: as for outcome 17
Time Frame: From date of randomization until 12 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 247 | 246
percentage of participants | 26.1 [20.7 to 31.9] | 11.7 [7.7 to 16.5]

20. Secondary Outcome: APF12 in PD-L1 TC >= 50% LREM Analysis Set
Description: as for outcome 17
Time Frame: From date of randomization until 12 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 207 | 199
percentage of participants | 26.5 [20.5 to 32.8] | 14.5 [9.6 to 20.4]

21. Secondary Outcome: Time From Randomization to Second Progression (PFS2)
Description: PFS2 was defined as the time from the date of randomization to the earliest of the progression events defined according to local clinical practice (subsequent to that used for the primary variable PFS) or death (i.e., date of PFS2 event or censoring - date of randomization + 1). PFS2 was calculated using the Kaplan-Meier technique.
Time Frame: Tumor assessments (per RECIST 1.1) until confirmed objective disease progression. Disease then assessed as per local practice until 2nd progression or death (up to a maximum of approximately 69 months)
Population: The FAS included all randomized participants who had PD-L1 expression TC >= 25% with the VENTANA PD-L1 (SP263) assay.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 335 | 334
months | 11.3 [9.8 to 12.7] | 9.3 [8.1 to 10.7]

22. Secondary Outcome: PFS2 in PD-L1 TC >= 25% LREM Analysis Set
Description: as for outcome 21
Time Frame: as for outcome 21
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 278 | 271
months | 11.8 [10.1 to 12.9] | 10.9 [9.3 to 13.1]

23. Secondary Outcome: PFS2 in PD-L1 TC >= 50% Analysis Set
Description: as for outcome 21
Time Frame: as for outcome 21
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 247 | 246
months | 11.3 [9.7 to 12.9] | 8.8 [8.0 to 10.9]

24. Secondary Outcome: PFS2 in PD-L1 TC >= 50% LREM Analysis Set
Description: as for outcome 21
Time Frame: as for outcome 21
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 207 | 199
months | 12.0 [10.1 to 13.8] | 10.9 [8.8 to 13.1]

25. Secondary Outcome: OS at 18 Months
Description: OS was defined as the time from the date of randomization until death due to any cause. Any participant not known to have died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive. The percentage of participants alive at 18 months were defined as the Kaplan-Meier estimate of OS at 18 months.
Time Frame: From date of randomization till 18 months.
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 335 | 334
percentage of participants | 42.5 [37.1 to 47.7] | 34.2 [29.0 to 39.4]

26. Secondary Outcome: OS at 18 Months in PD-L1 TC > = 25% LREM Analysis Set
Description: as for outcome 25
Time Frame: From date of randomization till 18 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 278 | 271
percentage of participants | 43.0 [37.1 to 48.8] | 41.4 [35.4 to 47.4]

27. Secondary Outcome: OS at 18 Months in PD-L1 TC >= 50% Analysis Set
Description: as for outcome 25
Time Frame: From date of randomization till 18 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 247 | 246
percentage of participants | 43.2 [36.9 to 49.3] | 34.9 [28.8 to 41.0]

28. Secondary Outcome: OS at 18 Months in PD-L1 TC >= 50% LREM Analysis Set
Description: as for outcome 25
Time Frame: From date of randomization till 18 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 207 | 199
percentage of participants | 44.3 [37.4 to 51.0] | 42.2 [35.2 to 49.1]

29. Secondary Outcome: OS at 24 Months
Description: OS was defined as the time from the date of randomization until death due to any cause. Any participant not known to have died at the time of analysis was censored based on the last recorded date on which the participant was known to be alive. The percentage of participants alive at 24 months were defined as the Kaplan-Meier estimate of OS at 24 months.
Time Frame: From date of randomization till 24 months
Population: The FAS included all randomized participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 335 | 334
percentage of participants | 34.6 [29.5 to 39.7] | 27.2 [22.4 to 32.1]

30. Secondary Outcome: OS at 24 Months in PD-L1 TC > = 25% LREM Analysis Set
Description: as for outcome 29
Time Frame: From date of randomization till 24 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 278 | 271
percentage of participants | 34.7 [29.1 to 40.3] | 32.8 [27.2 to 38.6]

31. Secondary Outcome: OS at 24 Months in PD-L1 TC >= 50% Analysis Set
Description: as for outcome 29
Time Frame: From date of randomization till 24 months
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 247 | 246
percentage of participants | 37.0 [31.0 to 43.1] | 27.0 [21.5 to 32.8]

32. Secondary Outcome: OS at 24 Months in PD-L1 TC >= 50% LREM Analysis Set
Description: as for outcome 29
Time Frame: From date of randomization till 24 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 207 | 199
percentage of participants | 36.9 [30.3 to 43.5] | 32.6 [26.1 to 39.3]

33. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) 30-Item Core Quality of Life Questionnaire Version 3 (QLQ-C30)
Description: The EORTC QLQ-C30 consisted of 30 questions that were combined to produce 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea/vomiting), 5 individual items (dyspnea, insomnia, appetite loss, constipation, and diarrhea), and a global measure of health status. The EORTC QLQ-C30 was scored according to the EORTC QLQ-C30 scoring manual. An outcome variable consisted of a score from 0 to 100. Higher scores on the global health status and functioning scales indicate better health status/function, but higher scores on symptom scales/items represent greater symptom severity. Baseline was defined as the last non-missing assessment prior to randomization. The mixed model repeated measures (MMRM) analysis of EORTC QLQ-C30 considered all data from baseline to PD or 12 months.
Time Frame: Baseline and 12 months
Population: The FAS included all randomized participants.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 268 | 249
scores on a scale
  Global health status | -0.7 (1.19) | -7.4 (1.27)
  Physical functioning | -3.3 (1.23) | -6.1 (1.30)
  Fatigue | 1.4 (1.33) | 7.2 (1.43)
  Appetite loss | -1.1 (1.39) | 9.1 (1.50)

34. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 in PD-L1 TC >= 25% LREM Analysis Set
Description: The EORTC QLQ-C30 consisted of 30 questions that were combined to produce 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea/vomiting), 5 individual items (dyspnea, insomnia, appetite loss, constipation, and diarrhea), and a global measure of health status. The EORTC QLQ-C30 was scored according to the EORTC QLQ-C30 scoring manual. An outcome variable consisted of a score from 0 to 100. Higher scores on the global health status and functioning scales indicate better health status/function, but higher scores on symptom scales/items represent greater symptom severity. Baseline was defined as the last non-missing assessment prior to randomization. The MMRM analysis of EORTC QLQ-C30 considered all data from baseline to PD or 12 months.
Time Frame: Baseline and 12 months
Population: The PD-L1 TC >= 25% LREM analysis set included participants identified by a prognostic model developed by AstraZeneca as having LREM. Only data from the participants analyzed were reported.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 236 | 208
scores on a scale
  Global health status | -1.4 (1.23) | -7.3 (1.31)
  Physical functioning | -3.9 (1.22) | -6.0 (1.29)
  Fatigue | 2.2 (1.33) | 7.7 (1.42)
  Appetite loss | -0.2 (1.43) | 9.8 (1.52)

35. Secondary Outcome: Time to Deterioration of EORTC QLQ-C30
Description: Time to symptom deterioration was defined as the time from the date of randomization until the date if the first clinically meaningful deterioration (a decrease in the function scales or the global health status/ health-related quality of life [HRQoL] from baseline of ≥10) that was confirmed at a subsequent visit or death in the absence of a clinically meaningful symptom deterioration, regardless of whether the participant withdraws from the study treatment or received another anticancer therapy prior to symptom deterioration. The EORTC QLQ-C30 consisted of 30 questions that were combined to produce 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea/vomiting), 5 individual items (dyspnea, insomnia, appetite loss, constipation, and diarrhea), and a global measure of health status. The EORTC QLQ-C30 was scored according to the EORTC QLQ-C30 scoring manual.
Time Frame: From randomization until date of first symptom deterioration that is confirmed, assessed up to a maximum of approximately 69 months (DCO 27 October 2022)
Population: The FAS included all randomized participants. Only data from the participants analyzed were reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 292 | 291
months
  Global health status: number analyzed (Participants) | 290 | 288
  Global health status | 7.3 [5.5 to 9.1] | 3.8 [3.6 to 5.5]
  Physical functioning | 7.4 [5.6 to 9.8] | 3.8 [3.6 to 5.2]
  Appetite loss: number analyzed (Participants) | 290 | 284
  Appetite loss | 9.2 [7.3 to 11.4] | 3.6 [2.3 to 3.8]
  Fatigue: number analyzed (Participants) | 290 | 289
  Fatigue | 4.9 [3.7 to 7.0] | 1.8 [1.6 to 2.6]

36. Secondary Outcome: Time to Deterioration of EORTC QLQ-C30 in PD-L1 TC >= 25% LREM Analysis Set
Description: Time to symptom deterioration was defined as the time from the date of randomization until the date if the first clinically meaningful deterioration a decrease in the function scales or the global health status/ HRQoL from baseline of ≥10) that was confirmed at a subsequent visit or death (by any cause) in the absence of a clinically meaningful symptom deterioration, regardless of whether the participant withdraws from the study treatment or received another anticancer therapy prior to symptom deterioration. The EORTC QLQ-C30 consisted of 30 questions that were combined to produce 5 functional scales (physical, role, cognitive, emotional, and social), 3 symptom scales (fatigue, pain, and nausea/vomiting), 5 individual items (dyspnea, insomnia, appetite loss, constipation, and diarrhea), and a global measure of health status. The EORTC QLQ-C30 was scored according to the EORTC QLQ-C30 scoring manual.
Time Frame: as for outcome 35
Population: as for outcome 34
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 253 | 239
months
  Global health status: number analyzed (Participants) | 250 | 238
  Global health status | 7.4 [5.6 to 9.2] | 5.5 [3.7 to 6.5]
  Physical functioning | 7.4 [5.6 to 10.1] | 4.7 [3.7 to 5.8]
  Appetite loss: number analyzed (Participants) | 251 | 233
  Appetite loss | 9.3 [7.3 to 11.6] | 3.7 [2.6 to 5.0]
  Fatigue: number analyzed (Participants) | 251 | 237
  Fatigue | 5.5 [3.8 to 7.4] | 1.8 [1.6 to 3.3]

37. Secondary Outcome: Change From Baseline in EORTC 13-Item Lung Cancer Quality of Life Questionnaire (QLQ-LC13)
Description: The QLQ-LC13 is a lung cancer specific module from the EORTC for lung cancer that comprised of 13 questions to assess lung cancer symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related side-effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and pain medication. An outcome variable consisted of a score from 0 to 100. Higher scores on symptom scales represent greater symptom severity. Baseline was defined as the last non-missing assessment prior to randomization. The MMRM analysis of EORTC QLQ-LC13 considered all data from baseline to PD or 12 months.
Time Frame: Baseline and 12 months
Population: The FAS included all randomized participants. Only data from the participants analyzed were reported.
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 274 | 259
scores on a scale
  Cough | -6.4 (1.30) | -7.9 (1.41)
  Dyspnea | 2.4 (1.24) | 4.1 (1.32)
  Chest pain | -1.0 (1.26) | -0.2 (1.37)

38. Secondary Outcome: Change From Baseline in EORTC QLQ-LC13 in PD-L1 TC >= 25% LREM Analysis Set
Description: as for outcome 37
Time Frame: Baseline and 12 months
Population: as for outcome 34
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 238 | 216
scores on a scale
  Cough | -6.6 (1.38) | -8.6 (1.48)
  Dyspnea | 2.9 (1.28) | 3.9 (1.35)
  Chest pain | -0.7 (1.30) | -1.0 (1.40)

39. Secondary Outcome: Time to Deterioration of EORTC QLQ-LC13
Description: Time to symptom deterioration was defined as the time from the date of randomization until the date if the first clinically meaningful symptom deterioration a decrease in the function scales or the global health status/ HRQoL from baseline of ≥10) that was confirmed at a subsequent visit or death (by any cause) in the absence of a clinically meaningful symptom deterioration, regardless of whether the participant withdraws from the study treatment or received another anticancer therapy prior to symptom deterioration. The QLQ-LC13 is a lung cancer specific module from the EORTC for lung cancer that comprised of 13 questions to assess lung cancer symptoms (cough, hemoptysis, dyspnea, and site-specific pain), treatment-related side-effects (sore mouth, dysphagia, peripheral neuropathy, and alopecia), and pain medication.
Time Frame: From randomization until date of first symptom deterioration that is confirmed, assessed up to maximum of approximately 69 months (DCO 27 October 2022)
Population: The FAS included all randomized participants. Only data from the participants analyzed were reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 284 | 281
months
  Cough: number analyzed (Participants) | 276 | 272
  Cough | 7.5 [6.4 to 10.1] | 6.6 [5.6 to 8.2]
  Dyspnea | 2.8 [1.9 to 4.6] | 3.6 [2.4 to 3.8]
  Chest pain: number analyzed (Participants) | 279 | 278
  Chest pain | 9.0 [6.3 to 11.9] | 6.4 [4.6 to 7.2]

40. Secondary Outcome: Time to Deterioration of EORTC QLQ-LC13 in PD-L1 TC >= 25% LREM Analysis Set
Description: as for outcome 39
Time Frame: as for outcome 39
Population: as for outcome 34
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 246 | 233
months
  Cough: number analyzed (Participants) | 239 | 225
  Cough | 9.2 [6.4 to 12.3] | 8.2 [6.4 to 11.1]
  Dyspnea | 3.6 [2.0 to 4.7] | 3.6 [2.4 to 3.8]
  Chest pain: number analyzed (Participants) | 242 | 231
  Chest pain | 9.8 [6.4 to 12.6] | 6.6 [5.8 to 9.2]

41. Secondary Outcome: Number of Participants With Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: ECOG performance status was assessed at the times specified based on the following and scored as 0: fully active: able to carry out all usual activities without restrictions. 1: Restricted in strenuous activity, but ambulatory and able to carry out any work activities; up and about more than 50% of waking hours. 3: Capable of only limited self-care; confined to bed or chair more than 50% of waking hours. 4: Completely disabled; unable to carry out any self-care and totally confined to bed or chair and 5: death. Data for only participants with restricted activity has been reported.
Time Frame: From Baseline and until follow-up period of 57 months
Population: The FAS included all randomized participants.
Measure: Number; unit: number of participants
Groups:
- Platinum-based SoC: Participants received 1 of the following IV infusion treatment combination platinum-based SoC as per Investigator's choice on Day 1 of each 21-day cycle for 4 to 6 cycles or until documented PD or until specific treatment discontinuation criteria were met.
  1. Paclitaxel 175 mg/m^2 and carboplatin AUC 5 or 6 via IV infusions.
  2. Gemcitabine 1000 or 1250 mg/m^2 and cisplatin 75 or 80 mg/m^2.
  3. Gemcitabine 1000 or 1250 mg/m^2 and carboplatin AUC 5 or 6 via infusions (for squamous participants).
  4. Pemetrexed 500 mg/m^2 and cisplatin 75 mg/m^2 (for non-squamous participants; pemetrexed maintenance dose was permitted).
  5. Pemetrexed 500 mg/m^2 and carboplatin AUC 5 or 6 via IV infusions (for non-squamous participants; pemetrexed maintenance dose was permitted).
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 335 | 334
number of participants
  Restricted activity, Baseline | 267 | 255
  Restricted activity, Follow-up Month 57 | 0 | 2

42. Secondary Outcome: Number of Participants With ECOG Performance Status in PD-L1 TC >=25% LREM Analysis Set
Description: as for outcome 41
Time Frame: From Baseline and until follow-up period of 57 months
Population: as for outcome 2
Measure: Number; unit: number of participants
Arm/Group | Durvalumab | Platinum-based SoC
Number analyzed (Participants) | 278 | 271
number of participants
  Restricted activity, Baseline | 221 | 203
  Restricted activity, Follow-up Month 57 | 0 | 2

43. Secondary Outcome: Percentage of Participants With Antidrug Antibody (ADA) Response to Durvalumab
Description: Treatment-emergent ADA positive was defined as either treatment-induced or treatment-boosted ADA. Treatment-boosted ADA was defined as a baseline positive ADA titer that was boosted to a 4-fold or higher-level following study drug administration. Persistently positive was defined as positive at least 2 post-baseline assessments with at least 16 weeks between the first and last positive assessment or positive at last post-baseline assessment. Transiently positive was defined as having at least 1 post-baseline ADA positive assessment and not fulfilling the conditions of persistently positive.
Time Frame: Up to 24 weeks
Population: The ADA evaluable analysis set included all participants in the safety analysis set who had a non-missing baseline ADA and at least 1 non-missing post-baseline ADA result.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 236
percentage of participants
  Treatment-emergent ADA positive | 0.8
  Treatment-boosted ADA | 0.4
  Persistently positive | 0
  Transiently positive | 0.8

44. Secondary Outcome: Percentage of Participants With ADA Response to Durvalumab in LREM Analysis Set
Description: as for outcome 43
Time Frame: Up to 24 weeks
Population: The ADA evaluable LREM analysis set included all participants in the safety analysis set who had a non-missing baseline ADA and at least 1 non-missing post-baseline ADA result, and identified by a prognostic model developed by AstraZeneca as having LREM.
Measure: Number; unit: percentage of participants
Arm/Group | Durvalumab
Number analyzed (Participants) | 208
percentage of participants
  Treatment-emergent ADA positive | 1.0
  Treatment-boosted ADA | 0.5
  Persistently positive | 0
  Transiently positive | 1.0

ADVERSE EVENTS:
Time Frame: From first administration of study treatment up to 90 days after the last dose of durvalumab or 30 days after last dose of platinum based SoC or date of initiation of the first subsequent therapy, whichever occurs first, for approximately 69 months.
Description: The Safety analysis set included all participants who received at least 1 dose of study treatment. All-cause mortality was in FAS analysis set.
Arm/Group | Durvalumab | Platinum-based SoC
All-Cause Mortality (participants affected / at risk) | 274/335 | 277/334
Serious Adverse Events (participants affected / at risk) | 132/335 | 104/327
Other Adverse Events (participants affected / at risk) | 271/335 | 294/327
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=335) | Platinum-based SoC (N=327)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Leukaemoid reaction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 2 (2)
Ileus (Gastrointestinal disorders) | 3 (3) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Asthenia (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 7 (7) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 4 (4)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 3 (3) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1)
Immune-mediated hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Liver injury (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Complicated appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Empyema (Infections and infestations) | 1 (3) | 1 (1)
Gastroenteritis shigella (Infections and infestations) | 1 (1) | 0 (0)
Myelosuppression (Blood and lymphatic system disorders) | 1 (1) | 14 (16)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Infectious pleural effusion (Infections and infestations) | 0 (0) | 1 (1)
Infusion site cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Lung abscess (Infections and infestations) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 19 (20)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Pneumonia (Infections and infestations) | 26 (33) | 17 (18)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 2 (2)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Nervous system injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood bilirubin increased (Investigations) | 2 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Coagulation time abnormal (Investigations) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1)
Neutrophil count increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 8 (9)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 0 (0) | 2 (2)
White blood cell count increased (Investigations) | 1 (1) | 0 (0)
Cachexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Immune-mediated myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to heart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bell's palsy (Nervous system disorders) | 0 (0) | 1 (1)
Brain oedema (Nervous system disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral artery embolism (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 4 (4) | 1 (2)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0)
Demyelination (Nervous system disorders) | 1 (1) | 0 (0)
Diplegia (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Immune-mediated encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Noninfective encephalitis (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's disease (Nervous system disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 4 (4) | 0 (0)
Completed suicide (Psychiatric disorders) | 2 (2) | 0 (0)
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (3) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Calculus prostatic (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Orchitis noninfective (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 4 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 4 (4)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 1 (1) | 0 (0)
Ventricular pre-excitation (Cardiac disorders) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 1 (1)
Deafness neurosensory (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Peripheral embolism (Vascular disorders) | 0 (0) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 0 (0) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durvalumab (N=335) | Platinum-based SoC (N=327)
Nausea (Gastrointestinal disorders) | 28 (29) | 107 (200)
Leukopenia (Blood and lymphatic system disorders) | 1 (15) | 51 (135)
Vomiting (Gastrointestinal disorders) | 17 (19) | 59 (97)
Asthenia (General disorders) | 37 (37) | 39 (66)
Fatigue (General disorders) | 22 (26) | 30 (38)
Non-cardiac chest pain (General disorders) | 17 (19) | 9 (9)
Pyrexia (General disorders) | 46 (82) | 25 (33)
Hepatic function abnormal (Hepatobiliary disorders) | 23 (29) | 17 (25)
Anaemia (Blood and lymphatic system disorders) | 81 (111) | 168 (266)
Neutropenia (Blood and lymphatic system disorders) | 4 (8) | 54 (134)
Pneumonia (Infections and infestations) | 27 (27) | 12 (12)
Thrombocytopenia (Blood and lymphatic system disorders) | 6 (10) | 34 (67)
Upper respiratory tract infection (Infections and infestations) | 33 (55) | 20 (22)
Alanine aminotransferase increased (Investigations) | 29 (45) | 45 (75)
Amylase increased (Investigations) | 21 (23) | 7 (8)
Aspartate aminotransferase increased (Investigations) | 27 (33) | 38 (62)
Gamma-glutamyltransferase increased (Investigations) | 15 (19) | 19 (24)
Haemoglobin decreased (Investigations) | 8 (13) | 17 (23)
Neutrophil count decreased (Investigations) | 9 (16) | 85 (251)
Platelet count decreased (Investigations) | 15 (25) | 56 (129)
Weight decreased (Investigations) | 46 (50) | 26 (26)
Weight increased (Investigations) | 21 (24) | 9 (11)
White blood cell count decreased (Investigations) | 13 (22) | 84 (291)
Decreased appetite (Metabolism and nutrition disorders) | 66 (80) | 94 (178)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 37 (50) | 18 (21)
Hypokalaemia (Metabolism and nutrition disorders) | 24 (40) | 26 (29)
Hyponatraemia (Metabolism and nutrition disorders) | 29 (33) | 24 (27)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 17 (17) | 4 (5)
Dizziness (Nervous system disorders) | 15 (16) | 21 (25)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 18 (18)
Insomnia (Psychiatric disorders) | 24 (27) | 24 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 29 (33) | 16 (17)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 19 (28) | 12 (12)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 9 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 42 (42)
Pruritus (Skin and subcutaneous tissue disorders) | 18 (18) | 6 (10)
Rash (Skin and subcutaneous tissue disorders) | 29 (32) | 7 (8)
Hypertension (Vascular disorders) | 20 (24) | 10 (12)
Hyperthyroidism (Endocrine disorders) | 24 (27) | 1 (1)
Hypothyroidism (Endocrine disorders) | 50 (85) | 2 (2)
Constipation (Gastrointestinal disorders) | 32 (36) | 57 (85)
Diarrhoea (Gastrointestinal disorders) | 23 (34) | 26 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/62/NCT03003962/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/62/NCT03003962/SAP_001.pdf